CLINICAL TRIAL: NCT04023396
Title: A Phase 2b, Open-label, Efficacy and Safety Study of ABX464 as Maintenance Therapy in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Efficacy and Safety Study of ABX464 as Maintenance Therapy in Patients With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX464-104
Record Dates: First submitted 2019-07-05; First posted 2019-07-17 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis
Keywords: moderate to severe ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: open-label, follow-up study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABX464 50mg (Experimental): All subjects will receive ABX464 administered at 50 mg o.d for an overall period of 96 weeks.
  Interventions: Drug: ABX464

INTERVENTIONS:
Drug: ABX464 — ABX464
  All subjects will receive ABX464 administered at 50 mg o.d for an overall period of 96 weeks.
  Other Names: Obefazimod

SUMMARY:
A phase 2b study to evaluate the long-term efficacy and safety study of ABX464 50mg as maintenance therapy in patients with moderate to severe Ulcerative Colitis.

DETAILED DESCRIPTION:
This study is an open-label study aiming at evaluating the long-term safety and the efficacy profile of ABX464 given once a day (o.d) at 50 mg in subjects who have been previously enrolled in the ABX464-103 clinical study (induction study) and who are willing to continue their treatment. All subjects will receive ABX464 given at 50mg o.d regardless of their previous treatment and dose received in the ABX464-103 study (i.e. ABX464 100mg, ABX464 50mg, ABX464 25mg or Placebo). The enrolment in this follow-up study will be based on the willingness of the subject to carry on his/her participation. Subjects will be treated with ABX464 for an overall period of 48 weeks. Subjects will be followed up on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the 16-week induction treatment period (ABX464-103);
* Patients are able and willing to comply with study visits and procedures as per protocol;
* Patients should understand, sign and date the written voluntary informed consent form prior to any protocol-specific procedures are performed;
* Patients should be affiliated to a social security regimen (for French sites only);
* Females and males receiving the study treatment (potentially in combination with immunosuppressant) and their partners must agree to use a highly effective contraceptive method during the study and for 6 months (180 days) after end of study or early termination. Contraception should be in place at least 2 weeks prior to screening. Women must be surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy) or in the postmenopausal state (no menses for 12 months without an alternative medical cause) or if of childbearing potential must use a highly effective contraceptive method. Women of childbearing potential (WOCBP) will enter the study after confirmed menstrual period and a negative pregnancy test. Highly effective methods of contraception include true abstinence, intrauterine device (IUD) or hormonal contraception aiming at inhibition of ovulation, intrauterine hormone releasing system, bilateral tubal ligation, vasectomized partner. True abstinence is defined when this is in line with the preferred and usual lifestyle of the patient. In each case of delayed menstrual period (over one month between menstruations) confirmation of absence of pregnancy is required. This recommendation also applies to WOCBP with infrequent or irregular menstrual cycle. Female and male patients must not be planning pregnancy during the trial and for 6 months post completion of their participation in the trial. In addition, male patients should use condom during the trial and for 6 months (180 days) post completion of their participation in the study. Male patients must not donate sperm as long as contraception is required.

Criteria that should be met by patients at week 48 to be eligible for 48 additional weeks of study treatment.

* Patients should be in clinical response. Clinical response is defined as: a reduction in Modified Mayo Score ≥ 2 points and ≥ 30 % from baseline (induction) with an accompanying decrease in rectal bleeding sub-score ≥ 1 point or absolute rectal bleeding sub-score ≤ 1 point.
* Patients able and willing to continue the study treatment and who are compliant with study visits and procedures and who signed the update of the written voluntary informed consent.

Exclusion Criteria:

* Patients who had major protocol deviation(s) in the induction study;
* Patients who permanently discontinued study the treatment in induction study (ABX464-103) because of an adverse event (AE) regardless of relatedness to investigational product;
* Patients who have developed any major illness/condition or evidence of an unstable clinical condition (except UC) that, in the investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study;
* Patients with any other severe acute or chronic medical or psychiatric condition or laboratory or electrocardiogram (ECG) abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study;
* Patients who are participating or plan to participate in other investigational studies (other than induction study) during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Severine VERMEIRE, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (120):
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - AKH - Medizinische Universität Wien, Vienna
- Belarus (5):
  - Gomel Regional Clinical Hospital, Homyel
  - Minsk city diagnostic center, Minsk
  - Regional Clinical Hospital, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
  - Vitebsk regoinal clinical specialized center, Vitebsk
- Belgium (3):
  - AZ Sint-Lucas, Bruges
  - C. H. U. St-Pierre, Brussels
  - University Hospitals Leuven - campus Gasthuisberg, Leuven
- Canada (5):
  - Brandon Medical Arts Clinic, Brandon
  - South Edmonton Gastroenterology, Edmonton
  - LHSC - Victoria Hospital, London
  - The Ottawa Hospital - General Campus, Ottawa
  - Mount Sinai Hospital, Toronto
- Czechia (7):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - MUDr. GREGAR s.r.o., Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Kunčice
  - Nemocnice Na Bulovce, Prague
  - Thomayerova nemocnice, Prague
  - Nemocnice Slany, Slaný
- France (18):
  - CHU Amiens - Hopital Sud, Amiens
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU de Grenoble - Hôpital Nord, Grenoble
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - CHU Lille - Hôpital Claude Huriez, Lille
  - Hôpital Nord - CHU Marseille, Marseille
  - Hopital Saint Eloi, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - CHU Nice - Hôpital de l'Archet 2, Nice
  - CHU Reims - Hôpital Robert Debré, Reims
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg
  - Hopital Rangueil, Toulouse
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (10):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Florence-Nightingale-Krankenhaus-Diakonie Kaiserswerth, Düsseldorf
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Studiengesellschaft BSF Unternehmergesellschaft haftungsbeschraenkt, Halle
  - Universitaetsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover, Hanover
  - Johanna-Etienne-Krankenhaus, Neuss
  - Tumorzentrum Nordthueringen MVZ GmbH, Nordhausen
  - Dr. Tasso Bieler, Riesa
  - Universitaetsklinikum Ulm, Ulm
- Hungary (7):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
  - Vasutegeszsegugyi Kft. - Debreceni Egeszsegugyi Kozpont, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
- Italy (10):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - I.R.C.C.S Policlinico San Donato, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
- Poland (15):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne Plejady, Krakow
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Wojskowy Szpital Kliniczny w Lublinie, Lublin
  - Trialmed CRS, Piotrkow Trybunalski
  - Centrum Medyczne Grunwald, Poznan
  - KO-MED Centra Kliniczne Pulawy, Puławy
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Centrum Zdrowia MDM, Warsaw
  - Nzoz Vivamed, Warsaw
  - Centrum Zdrowia Tuchow Sp. z o.o., Wierzchosławice
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - LexMedica, Wroclaw
- Serbia (3):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - General Hospital Uzice, Užice
- Slovakia (5):
  - Alian s.r.o., Bardejov
  - Gastromedic, s.r.o., Nové Zámky
  - Gastro I, s.r.o., Prešov
  - Accout Center s.r.o., Šahy
  - Endomed, s.r.o., Vranov nad Topľou
- Slovenia (3):
  - General Hospital Celje, Celje
  - University Medical Centre Maribor, Maribor
  - General Hospital Murska Sobota, Murska Sobota
- Spain (4):
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Quironsalud Malaga, Málaga
- Ukraine (17):
  - CNE Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Central City Clinical Hospital Dept of Theraphy No. 2 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv
  - Communal Non-commercial Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - CI Kherson CCH, Kherson
  - Khmelnytska Regional Hospital, Khmelnytskyi
  - Communal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Lviv Regional Clinical Hospital D.Halytskyi Lviv NMU, Lviv
  - Ternopil University Hospital, Ternopil
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - CI City Clinical Hospital #6 Dept of Gastroenterology, Zaporizhzhia
  - CNCE "City Hospital 9" Zaporizhzhia CC, Zaporizhzhia
- United Kingdom (4):
  - Fairfield General Hospital, Bury
  - Guy's Hospital, London
  - University College London Hospitals, London
  - Nottingham University Hospitals Queen's Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermeire S, Nitcheu J, Gineste P, Flatres A, Santo J, Scherrer D, Peyrin-Biroulet L, Dulai PS, Danese S, Dubinsky M, Tilg H, Siegmund B, Hisamatsu T, Shan K, Rabbat CJ, Sands BE. Obefazimod in patients with moderate-to-severely active ulcerative colitis: efficacy and safety analysis from the 96-week open-label maintenance phase 2b study. J Crohns Colitis. 2025 May 8;19(5):jjaf074. doi: 10.1093/ecco-jcc/jjaf074. PMID 40417999
- [Derived] Vermeire S, Sands BE, Tilg H, Tulassay Z, Kempinski R, Danese S, Bunganic I, Nitcheu J, Santo J, Scherrer D, Biguenet S, Ehrlich HJ, Steens JM, Gineste P, Sandborn WJ. ABX464 (obefazimod) for moderate-to-severe, active ulcerative colitis: a phase 2b, double-blind, randomised, placebo-controlled induction trial and 48 week, open-label extension. Lancet Gastroenterol Hepatol. 2022 Nov;7(11):1024-1035. doi: 10.1016/S2468-1253(22)00233-3. Epub 2022 Sep 6. PMID 36075249

RESULTS

PARTICIPANT FLOW:
Groups:
- ABX464 50mg: All subjects will receive ABX464 administered at 50 mg o.d for an overall period of 96 weeks.
  ABX464: ABX464
  All subjects will receive ABX464 administered at 50 mg o.d for an overall period of 96 weeks.
Period: Overall Study
Arm/Group | ABX464 50mg
Started | 217
Completed | 164
Not Completed | 53
Not completed — Adverse Event | 16
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 14
Not completed — Pregnancy | 4
Not completed — Lack of Efficacy | 3
Not completed — Physician Decision | 4
Not completed — Other reason (e.g., Ukraine Crisis) | 10

BASELINE CHARACTERISTICS:
Population: Patients with moderate to severe UC who were previously enrolled in the ABX464 103 clinical study (induction study).
  All patients who completed the 16-week (± 4 days) induction treatment period (ABX464-103) were eligible for this maintenance study regardless of their clinical response.
  Enrolled patients in ABX464 104 clinical study were willing to continue treatment with ABX464 as long-term (maintenance) therapy of remission.
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (13.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 133
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hungary | 17
  Czechia | 12
  Ukraine | 30
  Spain | 1
  Canada | 5
  Austria | 7
  Belgium | 8
  Poland | 63
  Italy | 17
  Slovakia | 16
  Slovenia | 3
  France | 24
  Serbia | 5
  Germany | 9

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Clinical Remission at Week 48 Compared to Baseline of Induction Study (ABX464-103)
Description: Clinical remission (based on the Mayo scoring system) is defined as: a rectal bleeding sub-score = 0, and an endoscopy sub-score ≤1 (excluding friability), and at least 1-point decrease in stool frequency sub-score from baseline to achieve a stool frequency sub-score ≤1
Time Frame: week 48
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
Participants | 119

2. Secondary Outcome: Proportion of Patients With Clinical Response at Weeks 48 and 96 Compared to Baseline of Induction Study
Description: Proportion of patients with clinical response at week 48 Clinical response is defined as: a reduction in Mayo Score ≥ 3 points and ≥ 30 % from baseline with an accompanying decrease in rectal bleeding sub-score ≥ 1 point or absolute rectal bleeding sub-score ≤ 1 point.
Time Frame: Weeks 48 and 96
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
Participants
  Week 48 | 177
  Week 96 | 158

3. Secondary Outcome: Endoscopic Improvement at Weeks 48 and 96
Description: Proportion of patients with endoscopic improvement at week 48 among all patients.
  Proportion of patients with endoscopic improvement at week 96 among all patients.
  Endoscopic improvement is defined as a Mayo endoscopic sub score of ≤1 (excluding friability).
Time Frame: week 48 and week 96
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
Participants
  Week 48 | 133
  Week 96 | 128

4. Secondary Outcome: Endoscopic Remission at Weeks 48 and 96
Description: Proportion of patients with endoscopic remission at week 48 among all patients. Proportion of patients with endoscopic remission at week 96 among all patients. Endoscopic remission is defined as a Mayo endoscopic sub score of 0.
Time Frame: week 48 and week 96
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
Participants
  Week 48 | 72
  Week 96 | 78

5. Secondary Outcome: Sustained Endoscopic Changes at Week 48 and Week 96
Description: Proportion of patients with sustained endoscopic changes at week 48 and 96. Sustained endoscopic changes is defined as the number of patients with endoscopic changes at week 48 among patients who had endoscopic changes during the Induction study (at week 8 or week 16 of study ABX464-103).
Time Frame: weeks 48 and 96
Population: At Week 8 of the induction study, endoscopic improvement was achieved by 70 patients; 16 patients achieved endoscopic remission
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
Participants
  Sustained endoscopic improvement at Week 48: number analyzed (Participants) | 70
  Sustained endoscopic improvement at Week 48 | 53
  Sustained endoscopic remission at Week 48: number analyzed (Participants) | 16
  Sustained endoscopic remission at Week 48 | 13
  Sustained endoscopic improvement at Week 96: number analyzed (Participants) | 70
  Sustained endoscopic improvement at Week 96 | 50
  Sustained endoscopic remission at Week 96: number analyzed (Participants) | 16
  Sustained endoscopic remission at Week 96 | 11

6. Secondary Outcome: Change in Modified Mayo Score and in Partial Modified Mayo Score
Description: Change in Modified Mayo Score (MMS) at weeks 48 and 96 and in partial Modified Mayo Score (pMMS)
  MMS is a composite score of UC disease activity calculated as the sum of the following 3 subscores:
  1. Stool frequency, scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding, scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic evaluation, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall MMS ranges from 0 to 9 where higher scores represent more severe disease.
  pMMS is a composite score of UC disease activity calculed as the sum of the following 2 subscores:
  1. Stool frequency, scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding, scored from 0 (no blood seen) to 3 (blood alone passed). The overall pMMS ranges from 0 to 6 where higher scores represent more severe disease.
Time Frame: From baseline to week 96
Population: Number of patients in the Full analysis set is 217; number analyzed in different rows correspond to number of patients analysed in the relevant week (lower than the overall number analyzed in FAS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
units on a scale
  MMS baseline ISB | 7.0 (1.07)
  MMS baseline BOLS: number analyzed (Participants) | 151
  MMS baseline BOLS | 4.0 (2.02)
  MMS Week 48: number analyzed (Participants) | 182
  MMS Week 48 | 1.8 (1.47)
  MMS Week 96: number analyzed (Participants) | 154
  MMS Week 96 | 1.5 (1.48)
  pMMS baseline ISB | 4.2 (1.01)
  pMMS baseline BOLS: number analyzed (Participants) | 214
  pMMS baseline BOLS | 1.8 (1.31)
  pMMS Week 4: number analyzed (Participants) | 214
  pMMS Week 4 | 1.4 (1.17)
  pMMS Week 8: number analyzed (Participants) | 208
  pMMS Week 8 | 1.4 (1.24)
  pMMS Week 12: number analyzed (Participants) | 203
  pMMS Week 12 | 1.3 (1.22)
  pMMS Week 16: number analyzed (Participants) | 200
  pMMS Week 16 | 1.3 (1.2)
  pMMS Week 20: number analyzed (Participants) | 196
  pMMS Week 20 | 1.2 (1.14)
  pMMS Week 24: number analyzed (Participants) | 192
  pMMS Week 24 | 1.1 (1.06)
  pMMS Week 28: number analyzed (Participants) | 191
  pMMS Week 28 | 1.1 (1.09)
  pMMS Week 32: number analyzed (Participants) | 189
  pMMS Week 32 | 1.0 (1.00)
  pMMS Week 36: number analyzed (Participants) | 188
  pMMS Week 36 | 1.0 (0.98)
  pMMS Week 40: number analyzed (Participants) | 185
  pMMS Week 40 | 0.9 (0.94)
  pMMS Week 44: number analyzed (Participants) | 182
  pMMS Week 44 | 0.9 (0.98)
  pMMS Week 48: number analyzed (Participants) | 184
  pMMS Week 48 | 0.8 (0.88)
  pMMS Week 60: number analyzed (Participants) | 175
  pMMS Week 60 | 0.7 (0.80)
  pMMS Week 72: number analyzed (Participants) | 170
  pMMS Week 72 | 0.7 (0.84)
  pMMS Week 84: number analyzed (Participants) | 169
  pMMS Week 84 | 0.7 (0.93)
  pMMS Week 96: number analyzed (Participants) | 165
  pMMS Week 96 | 0.7 (0.79)

7. Secondary Outcome: Stool Frequency Subscore
Description: Participants recorded stool frequency using a paper subject diary on a daily basis. The stool frequency subscore ranges from 0 to 3 according to the following scale:
  Score 0: Normal number of stools Score 1: 1 to 2 stools per day more than normal Score 2: 3 to 4 stools per day more than normal Score 3: 5 or more stools per day more than normal
Time Frame: From baseline to week 96
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
score on a scale
  Stool frequency - Baseline ISB | 2.6 (0.66)
  Stool frequency - Baseline BOLS: number analyzed (Participants) | 214
  Stool frequency - Baseline BOLS | 1.4 (0.94)
  Stool frequency - Week 4: number analyzed (Participants) | 214
  Stool frequency - Week 4 | 1.2 (0.89)
  Stool frequency - Week 8: number analyzed (Participants) | 209
  Stool frequency - Week 8 | 1.2 (0.93)
  Stool frequency - Week 12: number analyzed (Participants) | 203
  Stool frequency - Week 12 | 1.1 (0.93)
  Stool frequency - Week 16: number analyzed (Participants) | 202
  Stool frequency - Week 16 | 1.1 (0.93)
  Stool frequency - Week 20: number analyzed (Participants) | 198
  Stool frequency - Week 20 | 1.0 (0.92)
  Stool frequency - Week 24: number analyzed (Participants) | 193
  Stool frequency - Week 24 | 1.0 (0.83)
  Stool frequency - Week 28: number analyzed (Participants) | 192
  Stool frequency - Week 28 | 0.9 (0.87)
  Stool frequency - Week 32: number analyzed (Participants) | 190
  Stool frequency - Week 32 | 0.9 (0.78)
  Stool frequency - Week 36: number analyzed (Participants) | 189
  Stool frequency - Week 36 | 0.9 (0.82)
  Stool frequency - Week 40: number analyzed (Participants) | 185
  Stool frequency - Week 40 | 0.8 (0.8)
  Stool frequency - Week 44: number analyzed (Participants) | 182
  Stool frequency - Week 44 | 0.8 (0.8)
  Stool frequency - Week 48: number analyzed (Participants) | 184
  Stool frequency - Week 48 | 0.7 (0.79)
  Stool frequency - Week 60: number analyzed (Participants) | 176
  Stool frequency - Week 60 | 0.7 (0.73)
  Stool frequency - Week 72: number analyzed (Participants) | 170
  Stool frequency - Week 72 | 0.7 (0.76)
  Stool frequency - Week 84: number analyzed (Participants) | 169
  Stool frequency - Week 84 | 0.7 (0.77)
  Stool frequency - Week 96: number analyzed (Participants) | 165
  Stool frequency - Week 96 | 0.6 (0.73)

8. Secondary Outcome: Rectal Bleeding Score
Description: Participants recorded rectal bleeding in a paper subject diary on a daily basis. Rectal bleeding score is taken as the worst subscore of the three most recent scores within 7 days prior to the visit.
  The rectal bleeding subscore ranges from 0 to 3 according to the following scale:
  Score 0: No blood seen Score 1: Streaks of blood with stool less than half the time Score 2: Obvious blood with stool most of the time Score 3: Blood alone passed A lower score represents an improvement in rectal bleeding.
Time Frame: From baseline to week 96
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
score on a scale
  Rectal bleeding Score - Baseline ISB | 1.6 (0.72)
  Rectal bleeding Score - Baseline BOLS: number analyzed (Participants) | 214
  Rectal bleeding Score - Baseline BOLS | 0.4 (0.66)
  Rectal bleeding Score - Week 4: number analyzed (Participants) | 214
  Rectal bleeding Score - Week 4 | 0.2 (0.49)
  Rectal bleeding Score - Week 8: number analyzed (Participants) | 208
  Rectal bleeding Score - Week 8 | 0.2 (0.56)
  Rectal bleeding Score - Week 12: number analyzed (Participants) | 203
  Rectal bleeding Score - Week 12 | 0.2 (0.50)
  Rectal bleeding Score - Week 16: number analyzed (Participants) | 200
  Rectal bleeding Score - Week 16 | 0.2 (0.51)
  Rectal bleeding Score - Week 20: number analyzed (Participants) | 196
  Rectal bleeding Score - Week 20 | 0.2 (0.49)
  Rectal bleeding Score - Week 24: number analyzed (Participants) | 192
  Rectal bleeding Score - Week 24 | 0.2 (0.46)
  Rectal bleeding Score - Week 28: number analyzed (Participants) | 191
  Rectal bleeding Score - Week 28 | 0.1 (0.42)
  Rectal bleeding Score - Week 32: number analyzed (Participants) | 189
  Rectal bleeding Score - Week 32 | 0.1 (0.39)
  Rectal bleeding Score - Week 36: number analyzed (Participants) | 188
  Rectal bleeding Score - Week 36 | 0.1 (0.38)
  Rectal bleeding Score - Week 40: number analyzed (Participants) | 185
  Rectal bleeding Score - Week 40 | 0.1 (0.37)
  Rectal bleeding Score - Week 44: number analyzed (Participants) | 182
  Rectal bleeding Score - Week 44 | 0.1 (0.37)
  Rectal bleeding Score - Week 48: number analyzed (Participants) | 184
  Rectal bleeding Score - Week 48 | 0.0 (0.23)
  Rectal bleeding Score - Week 60: number analyzed (Participants) | 175
  Rectal bleeding Score - Week 60 | 0.0 (0.24)
  Rectal bleeding Score - Week 72: number analyzed (Participants) | 170
  Rectal bleeding Score - Week 72 | 0.0 (0.24)
  Rectal bleeding Score - Week 84: number analyzed (Participants) | 169
  Rectal bleeding Score - Week 84 | 0.1 (0.36)
  Rectal bleeding Score - Week 96: number analyzed (Participants) | 165
  Rectal bleeding Score - Week 96 | 0.0 (0.22)

9. Secondary Outcome: C-Reactive Protein
Description: Change to baseline in C-Reactive Protein levels
Time Frame: baseline, week 24, week 48
Population: Number of patients in the Full analysis set is 217; number analyzed in different rows correspond to number of patients analysed in the relevant week
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
mg/L
  Baseline BOLS: number analyzed (Participants) | 216
  Baseline BOLS | 6.66 (12.17)
  Week 24: number analyzed (Participants) | 191
  Week 24 | 5.07 (10.43)
  Week 48: number analyzed (Participants) | 183
  Week 48 | 5.01 (11.31)

10. Secondary Outcome: miRNA-124 Expression
Description: Change relative to baseline in miRNA-124 expression in rectal/sigmoidal biopsies at week 48 and in total blood at week 24 and week 48.
Time Frame: baseline, week 24 and week 48
Population: Absolute quantification (QuantaSoft Pro) of the miR-124 copy number was performed at baseline of the induction study, at week 48 and at week 96 by using droplet digital PCR technology on 115 whole blood samples and 240 rectal biopsy samples.
Measure: Mean (Standard Deviation); unit: copy number/cell
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
copy number/cell
  miR-124 - Rectal - Baseline | 0.00065 (0.00211)
  miR-124 - Rectal - Week 48 | 0.00255 (0.00252)
  miR-124 - Sigmoidal- Baseline | 0.00035 (0.00050)
  miR-124 - Sigmoidal- Week 48 | 0.00225 (0.00216)
  miR-124 - Blood- Baseline | 0.00000 (0.00000)
  miR-124 - Blood- Week 24 | 0.00011 (0.00015)
  miR-124 - Blood- Week 48 | 0.00013 (0.00026)

11. Secondary Outcome: Incidence and Description of Adverse Events
Description: Number and rate of all adverse events, causally-related adverse events, all serious adverse events and causally-related serious adverse events classified by severity.
  Incidence of treatment-emergent serious adverse events, hospitalizations, total inpatient days.
  Incidence of adverse events leading to investigational product discontinuation. Number of clinically significant laboratory abnormalities.
Time Frame: From baseline to week 96
Population: the safety analysis set (SAF) included all patients who had at least one dose of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg
Number analyzed (Participants) | 217
Participants
  AEs | 149
  TEAEs | 148
  Related TEAEs | 54
  SAEs | 18
  TESAEs | 18
  TEAEs leading to discontinuation of investigational product | 26
  TEAEs leading to study discontinuation | 17

ADVERSE EVENTS:
Time Frame: 96 weeks
Description: no difference
Arm/Group | ABX464 50mg
All-Cause Mortality (participants affected / at risk) | 1/217
Serious Adverse Events (participants affected / at risk) | 18/217
Other Adverse Events (participants affected / at risk) | 148/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 50mg (N=217)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Colon dysplasia (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Apendicitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneunomia (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Ischemic stroke (Nervous system disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 50mg (N=217)
COVID-19 (Infections and infestations) | 31 (34)
Nasopharyngitis (Infections and infestations) | 15 (23)
Upper respiratory tract infection (Infections and infestations) | 6 (7)
Pharyngitis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 3 (3)
Blood cholesterol increased (Investigations) | 8 (10)
C-reactive protein increased (Investigations) | 6 (7)
Low density lipoprotein increased (Investigations) | 5 (7)
Alanine aminotransferase increased (Investigations) | 4 (6)
Neutrophil count increased (Investigations) | 4 (4)
Thyroxine increased (Investigations) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Lipase increased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 3 (3)
SARS-CoV-2 test positive (Investigations) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 17 (20)
Abdominal pain (Gastrointestinal disorders) | 8 (10)
Nausea (Gastrointestinal disorders) | 8 (8)
Hemorrhoids (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 25 (35)
Vaccination complication (Injury, poisoning and procedural complications) | 5 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
Folate deficiency (Metabolism and nutrition disorders) | 6 (6)
Hypercholesterolemia (Metabolism and nutrition disorders) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3)
Fecal calprotectin increased (Investigations) | 10 (11)
Fatigue (General disorders) | 4 (4)
Pyrexia (General disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Palpitations (Cardiac disorders) | 3 (4)
Ear infection (Infections and infestations) | 3 (3)
Hypertension (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT04023396/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT04023396/SAP_001.pdf